CLINICAL TRIAL: NCT07254299
Title: Hypnosis to Improve Well-beings of Critically Ill Patients and Prevent Post-intensive Care Syndrome
Acronym: HypnoPICS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: COEN Matteo (Other)
Responsible Party: Sponsor-Investigator, COEN Matteo, Dr. med. PD. PhD, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-00369
Record Dates: First submitted 2025-11-14; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Post Intensive Care Syndrome (PICS)
Keywords: post intensive care syndrome; randomized controlled trail; hypnosis
MeSH Terms: conditions — postintensive care syndrome | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis group (Experimental): Participants in the intervention group will receive a hypnosis session on the day of discharge, a second session seven days post-discharge, and a third session on day 14 if they are still in the hospital. Trained professionals will conduct the hypnosis sessions following a standardized protocol, designed by the study team for critically ill patients.
  Interventions: Other: Hypnosis
- Control group (No Intervention): Participants in the control group will receive standard post-discharge care, which includes mobilization, nutrition, pain control, and family engagement and empowerment, without any hypnosis intervention.

INTERVENTIONS:
Other: Hypnosis — the hypnosis will be tailored to each patient. Key elements will include relaxation (to mitigate anxiety and stress and help the patient feel more comfortable, secure, and competent), reassociation techniques (to help the patient reconnect with their body, promoting a sense of embodiment and presence), and safe place (to introduce a safe and calming place to instill a sense of control and competence, aiding in emotional stabilization and fostering a sense of safety and well-being).
  Arms: Hypnosis group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of a hypnosis intervention in improving well-being at day 28 of an ICU stay. The main question it aims to answer is :

-Does Hypnosis intervention at ICU discharge and on day 7 and 14 on the wards if the patient remains in the hospital, improve wellbeing at 28 days ?

Researchers will compare discharged ICU patients who received standard post-discharge care to discharged ICU patients who received standard post-discharge care and hypnosis intervention on discharge and 7 and 14days after if they are still in the hospital, to see if hypnosis can improve their wellbeing.

Participants will receive a hypnosis session on the day of ICU discharge, a second session seven days post-discharge and a third session at day 14 if they are still in the hospital.

DETAILED DESCRIPTION:
Critically ill patients in the Intensive Care Unit (ICU) face numerous challenges both acutely and in the long term. These patients frequently experience acute pain and anxiety due to intubation and induced comas. Following their ICU discharge, they commonly report decreased well-being and quality of life. Additionally, up to 40% of critically ill patients develop post-intensive care syndrome (PICS), which includes mental, physical, and cognitive sequelae that can persist up to one year after discharge. Heavy sedation and medications necessary to manage pain and anxiety are known risk factors for PICS.

The current standard of care in the ICU includes mobilization and nutrition, pain control, and family engagement and empowerment. Furthermore, no other specific interventions are aimed at improving long-term outcomes and preventing PICS.

Several studies have explored using hypnosis to improve the acute care of ICU patients. For instance, a pain protocol that included hypnosis in burn patients hospitalized in the CHUV (Centre Hospitalier Universitaire Vaudois) resulted in reduced pain intensity, reduced opioid use, reduced anxiety, and better wound outcomes, all while lowering costs. A pilot study involving non-invasive ventilation patients showed that hypnosis could improve comfort, mask tolerance, and anxiety levels. Additionally, studies on relaxation therapy have indicated that electronic relaxation therapy is a promising, safe, and effective non-pharmacological solution to enhance overall comfort in alert and non-delirious ICU patients.

However, despite these efforts, there is a lack of efficient interventions specifically targeting the wellbeing of patients after an ICU stay and the prevention of PICS. Existing interventions, such as follow-up programs, rehabilitation, and psychological follow-up, have shown conflicting results. To date, no studies have specifically assessed the effect of hypnosis on the short and longer-term well-being of critically ill patients leaving the ICU and its possible effect on the prevention of PICS.

The investigators hypothesize that providing a hypnosis session at ICU discharge and followed by subsequent sessions on days 7 and 14 on the ward will improve well-being in the short term and reduce PICS symptoms at 3- and 6- months. The primary outcome will be the assessment of well-being at day 28 post-ICU discharge. Secondary outcomes will be anxiety, depression, PTSD, and quality of life at three and six months.

Hypothesis and primary objective The investigators hypothesize that providing intervention with hypnosis at ICU discharge and subsequent sessions on day 7 and 14 on the ward if the patient remains in the hospital will improve wellbeing at day 28 and reduce PICS symptoms at three and six months in critically ill patients.

Primary Objective:

The primary objective of this study is to evaluate the effectiveness of a hypnosis intervention in improving well-being at day 28 of an ICU stay.

Scale used for wellbeing:

* ESAS, total 90, each item on a 0-10 scale
* EQ-5D-5L

Secondary Objectives:

1. To assess the impact of a hypnosis intervention to improve PICS at 3 months and 6 months

   * Anxiety and depression: PHQ-9 et GAD-7
   * Post-traumatic stress disorder: PDI and IES-R scale
   * Quality of life: SF-12, EQ-5D-5L and WHODAS 2.0
   * Patient impression of change: PGIC
2. To evaluate patient immediate wellbeing after the hypnosis intervention. • ESAS before after the session in patients who will get the session

ELIGIBILITY:
Inclusion Criteria:

* On Mechanical Ventilation for at least 48 hours
* Able to give informed consent as documented by signature
* French speaking

Exclusion Criteria:

* Refusal of the patient
* Patient transferred from another ICU
* Patient is planned for a withdrawal of care or is actively dying
* Glasgow coma scale (GCS) <15 on ICU discharge
* Patient presenting with delirium (detected by CAM-ICU) on ICU discharge
* Patient hospitalized for brain injury
* Patient is in jail
* Patients already enrolled in the ongoing Nutriphyt trial
* Patient hospitalized for more than 28 days in the ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Wellbeing at day 28 post intensive care unit discharge | Day 28 post intensive care unit discharge
  ESAS scale (Edmonton Symptom Assessment System) with a range from 0 to 100. Higher scores means worse wellbeing.

SECONDARY OUTCOMES:
Immediate wellbeing following a hypnosis session | Day 1 (Day of discharge from ICU), day 7, day 14
  1) ESAS scale before and after the hypnosis session performed on Day 1 (ICU discharge), Day 7 and D14
  -The ESAS scale (Edmonton Symptom Assessment System) has a range from 0 to 100.
HADS | Day 28 post intensive care unit discharge, 3 months, 6 months post intensive care
  The HADS (Hospital Anxiety and Depression screening). The possible scores are: Anxiety subscale (HADS-A): 0-21 and Depression subscale (HADS-D): 0-21. Higher scores mean more depressive or anxiety symptoms.
IES-R (Impact of event Scale) | Day 28 post intensive care unit discharge, 3 months, 6 months post intensive care unit discharge. Higher score means more PTSD symptoms.
  Range: 0-88
SF-12 (Short Form 12-Item Health Survey) | Day 28 post intensive care unit discharge, 3 months, 6 months post intensive care unit discharge
  Main scores:
  * PCS-12 = Physical Component Summary
  * MCS-12 = Mental Component Summary
  Scoring / range:
  Items are combined using a scoring algorithm.
  Higher scores mean better quality of life.
EQ-5D-5L (Quality of life) | Day 28 post intensive care unit discharge, 3 months, 6 months post intensive care unit discharge
  Part 1) 5 dimensions: Mobility, Self-care, Usual activities, Pain/discomfort, Anxiety/depression. The 5-digit health state is converted (via country-specific value set) to an index value
  Part 2) EQ VAS (Visual Analog Scale). Patient rates their health today from 0 to 100.
  Higher scores mean better quality of life.
PGIC - Patient Global Impression of Change | Day 28 post intensive care unit discharge, 3 months, 6 months post intensive care unit discharge
  Single-item global rating of how much the patient feels their condition has changed since a reference time. Higher scores means improvement.
  Scoring / range: 1-7
PSQ - Patient Satisfaction Questionnaire (PSQ-18 short form) | Day 28 post intensive care unit discharge, 3 months, 6 months post intensive care unit discharge
  18 items total. Each item: 5-point Likert (1-5). Higher scores gives higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Wozniak, Medical Doctor, Principal Investigator — University Hospital, Geneva; Matteo Coen, MD, PHD, Principal Investigator — University Hospital, Geneva
Locations (2):
- Switzerland (2):
  - University Hospital of Geneva, Geneva
  - Hôpitaux Neuchâtelois, Neuchâtel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Schmidt B, Schneider J, Deffner T, Rosendahl J. Hypnotic suggestions of safety improve well-being in non-invasively ventilated patients in the intensive care unit. Intensive Care Med. 2021 Apr;47(4):485-486. doi: 10.1007/s00134-021-06364-8. Epub 2021 Feb 16. No abstract available. PMID 33590259
- [Result] Spiegel D, Cardena E. New uses of hypnosis in the treatment of posttraumatic stress disorder. J Clin Psychiatry. 1990 Oct;51 Suppl:39-43; discussion 44-6. PMID 2211565
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/12386494
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/17085255